CLINICAL TRIAL: NCT04826211
Title: Targeting the Future of Axillary Staging in Node Positive Breast Cancer Patients Receiving Primary Systemic Therapy. A Comparative Study Between Sentinel Node Biopsy vs PET/MRI.
Brief Title: Axillary Staging in Node Positive Breast Cancer Patients Receiving PST. SNB vs PET/MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Oreste Davide Gentilini, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNB vs PET/MRI 1
Record Dates: First submitted 2020-05-25; First posted 2021-04-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Female; Node-positive Breast Cancer; Sentinel Lymph Node
Keywords: primary systemic therapy; node positive breast cancer; surgery after primary systemic therapy; PET/MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Node positive BC patients undergoing PST (Experimental): Patients with breast cancer of any size with positive axillary nodes and candidates to PST will undergo PET/MRI both prior to PST and after PST before surgery
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — All included patients will undergo PET/MRI both prior to PST and prior to surgery. In order to analyze results the population will be divided into two groups: women with positive axillary lymph nodes after PST (Group 1) and women with negative axillary lymph nodes after PST (Group 2).

SUMMARY:
The management of axillary nodes in breast cancer patients is a highly debated and evolving field. To date, an increasing number of patients with positive lymph nodes receives primary systemic therapy (PST) prior to surgery leading to down-staging axillary nodes in about 40% of women. However, the available diagnostic methods have several limitations in properly evaluating the response after treatment both in the breast and in the nodes and might lead to either under or over-treatment in these patients. Fully integrated scanners capable of simultaneous acquisition of PET and MRI have now been developed, with the potential to combine the specificity obtained by the functional imaging of PET, with the superior sensitivity of MRI, to provide higher diagnostic accuracy.

It is expected that PET/MRI could better determine the response after PST to distinguish patients with negative versus patients with positive axillary nodes after medical treatment. As the excision of axillary nodes has mainly a staging purpose, the reliable identification of node negative patients might eventually spare women from unnecessary surgery. An accurate over-time and final imaging work-up might help choose the appropriate type of surgery according to the extent of nodal involvement: either SNB or complete axillary clearance.

DETAILED DESCRIPTION:
HYPOTHESIS: Hybrid PET/MRI might be a non-invasive, one-stage, operator-independent imaging modality to accurately define nodal status after PST, properly select type of surgical approach and might eventually lead to the omission of axillar surgery in some breast cancer patients showing complete imaging response.

AIMS: The primary endpoint is to compare the staging power between SNB (or lymphoadenectomy) vs PET/MRI in detecting axillary lymph node macro-metastases (>2 mm).Additionally the PET/MRI and A-US results will be confronted and ultimately related to pathology result, calculating the concordance rate in terms of positive vs negative nodes and number of positive nodes detected by each method. The staging power of both preoperative exams will be evaluated by considering how many times the results from PET/MRI or A-US could have indicated the most appropriate axillary treatment according to pathological findings.

EXPERIMENTAL DESIGN: Patients with breast cancer of any size with positive axillary nodes and candidates to PST will undergo PET/MRI prior to PST.

The study population will then be split into two groups:

* women with positive axillary lymph nodes after PST (Group 1, 60% of the total)
* women with negative axillary lymph nodes after PST (Group 2, 40% of the total).

A total of 110 women will guarantee two well-powered independent analysis. one for Group 1 (n=66; power>90%; Type I error rate of 0.05) and one for Group 2 (n=44; power>80%; Type I error rate of 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age > 18 years;
* Proven diagnosis of early BC of any size;
* Patients candidate to primary systemic therapy (PST);
* Positive axillary nodes at diagnosis, confirmed by either citology or histology confirmation. Patients with clear overt clinical and radiological nodal involvement might be enrolled as well without FNA or microhystology

Exclusion Criteria:

* inflammatory BC;
* pregnancy;
* contraindication to PET;
* distant metastases;
* no surgery after PST;
* contraindication to MRI;
* claustrophobia;
* allergy to the MR contrast agent;
* severe renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Axillary surgery vs PET/MRI. | Within 1 month after surgery results from axillary surgery will be available and compared to preoperative PET/MRI
  Results from SNB (Sentinel Node Biopsy), AD (Axillary Dissection) or any axillary surgery will be compared to results from preoperative PET/MRI.

SECONDARY OUTCOMES:
Staging power of PET/MRI will be compared to preoperative A-US (Axillary ultrasound) | At 12 months
  Results on the status of axillary nodes from preoperative A-US will be compared to results of preoperative PET/MRI.
Correlation between PET/MRI parameters and prognosis | At baseline and at 5 years
  Quantitative analysis of PET/MRI exams will allow to extract standard imaging biomarkers to be correlated with tumour clinical and pathological data. Image analysis will be carried out both at staging and at the end of PST.
  Functional parameters from PET image analysis include Standardized Uptake Value and Metabolic Tumor Volume.
  From breast MR images, the quantitative and semiquantitative data are related to DWI and DCE MR sequences. Specifically, from the so-called Time Intensity Curve (TIC) obtained from the dynamic DCE some parameters can be extracted, for example Time To Peak, Peak Enhancement Percentage, Signal Enhancement Ratio and Initial Enhancement Percentage. From DWI MR sequence Apparent Diffusion Coefficient map can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: GENTILINI, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taneja S, Jena A, Goel R, Sarin R, Kaul S. Simultaneous whole-body (1)(8)F-FDG PET-MRI in primary staging of breast cancer: a pilot study. Eur J Radiol. 2014 Dec;83(12):2231-2239. doi: 10.1016/j.ejrad.2014.09.008. Epub 2014 Sep 28. PMID 25282709
- [Background] Melsaether AN, Raad RA, Pujara AC, Ponzo FD, Pysarenko KM, Jhaveri K, Babb JS, Sigmund EE, Kim SG, Moy LA. Comparison of Whole-Body (18)F FDG PET/MR Imaging and Whole-Body (18)F FDG PET/CT in Terms of Lesion Detection and Radiation Dose in Patients with Breast Cancer. Radiology. 2016 Oct;281(1):193-202. doi: 10.1148/radiol.2016151155. Epub 2016 Mar 29. PMID 27023002
- [Background] Veronesi U, De Cicco C, Galimberti VE, Fernandez JR, Rotmensz N, Viale G, Spano G, Luini A, Intra M, Veronesi P, Berrettini A, Paganelli G. A comparative study on the value of FDG-PET and sentinel node biopsy to identify occult axillary metastases. Ann Oncol. 2007 Mar;18(3):473-8. doi: 10.1093/annonc/mdl425. Epub 2006 Dec 12. PMID 17164229
- [Background] Gentilini O, Veronesi U. Staging the Axilla in Early Breast Cancer: Will Imaging Replace Surgery? JAMA Oncol. 2015 Nov;1(8):1031-2. doi: 10.1001/jamaoncol.2015.2337. No abstract available. PMID 26291922
- [Background] van Nijnatten TJA, Goorts B, Voo S, de Boer M, Kooreman LFS, Heuts EM, Wildberger JE, Mottaghy FM, Lobbes MBI, Smidt ML. Added value of dedicated axillary hybrid 18F-FDG PET/MRI for improved axillary nodal staging in clinically node-positive breast cancer patients: a feasibility study. Eur J Nucl Med Mol Imaging. 2018 Feb;45(2):179-186. doi: 10.1007/s00259-017-3823-0. Epub 2017 Sep 14. PMID 28905091
- [Background] Heusch P, Nensa F, Schaarschmidt B, Sivanesapillai R, Beiderwellen K, Gomez B, Kohler J, Reis H, Ruhlmann V, Buchbender C. Diagnostic accuracy of whole-body PET/MRI and whole-body PET/CT for TNM staging in oncology. Eur J Nucl Med Mol Imaging. 2015 Jan;42(1):42-8. doi: 10.1007/s00259-014-2885-5. Epub 2014 Aug 12. PMID 25112399
- [Background] Stadnik TW, Everaert H, Makkat S, Sacre R, Lamote J, Bourgain C. Breast imaging. Preoperative breast cancer staging: comparison of USPIO-enhanced MR imaging and 18F-fluorodeoxyglucose (FDC) positron emission tomography (PET) imaging for axillary lymph node staging--initial findings. Eur Radiol. 2006 Oct;16(10):2153-60. doi: 10.1007/s00330-006-0276-4. Epub 2006 May 3. PMID 16670863